CLINICAL TRIAL: NCT03160404
Title: The Effects of Zolpidem Compared With Exercise on Chronic Insomnia
Brief Title: Zolpidem or Exercise for Insomnia?
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Giselle Soares Passos, Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.986.600
Record Dates: First submitted 2017-05-04; First posted 2017-05-19 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Chronic Insomnia
Keywords: Exercise; Zolpidem; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity | interventions — Zolpidem; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXERCISE (Experimental): Aerobic exercise (50% Reserve heart hate), 50 minutes, 3 times/week, during 6 weeks.
  Interventions: Behavioral: Exercise
- ZOLPIDEM (Active Comparator): 10 mg/night during 6 weeks
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: Zolpidem — The ZOLPIDEM group will be treated with zolpidem 10mg/night
  Arms: ZOLPIDEM
Behavioral: Exercise — The EXERCISE group will participate in an aerobic exercise program, performed in intensity relative to 50% of reserve heart rate, on a treadmill.
  Arms: EXERCISE

SUMMARY:
Introduction: The prevalence of chronic insomnia in the general population is between 10 and 15%. The therapy commonly prescribed for its treatment is pharmacological, however, there are several non-pharmacological alternatives being studied, among them physical exercise. Although some studies have described the effect of exercise on sleep in insomnia, there are no studies comparing exercise and drugs in the treatment of chronic insomnia, or its effect as coadjuvant therapy.

Objective: To compare the acute and chronic effects of aerobic exercise and zolpidem on sleep quality, mood and quality of life in patients with chronic insomnia.

Material and Methods: 30 patients with chronic insomnia will be randomly assigned into two groups: EXERCISE (n=15) or ZOLPIDEM (n=15). The patients of EXERCISE group will be included in an aerobic exercise program, performed in 50% of reserve heart rate, on a treadmill (50 minutes, 3 times/week), during 6 weeks. The ZOLPIDEM group will be treated with zolpidem (10mg/night) during 6 weeks. Polysomnography, actigraphy, sleep diary and questionnaires will be used the evaluate sleep pattern. Mood and quality of life will be investigated by POMS and SF-36 questionnaires.

Hypothesis: Considering previous studies have demonstrated positive effects of aerobic exercise in the insomnia symptoms, the hypothesis of this study is that aerobic exercise, performed at moderate intensity, can control the symptoms of chronic insomnia similarly to pharmacological therapy.

ELIGIBILITY:
Inclusion criteria:

* age 30 -60 years;
* clinical diagnosis of chronic insomnia according to the DSM-V;
* insomnia complaint at least 3 times a week for at least 3 months;
* be physically inactive (exercise less than 2 times a week).

Exclusion criteria:

* evidence that insomnia is directly related to medical conditions or side effects of medications;
* obstructive sleep apnea syndrome;
* ECG abnormalities that prevent physical exercise or use of beta-blockers;
* uncontrolled clinical diseases (diabetes, hypertension, cardiovascular, neurological or renal diseases);
* use or history of abuse of alcohol or psychoactive substances);
* use of sleeping pills> 2 times a week;
* shift workers.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline polysomographic sleep recording to first night and 6 weeks | baseline, first night, week 6
  Polysomnografic recording include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram. Measurements of air flow (oral and nasal), respiratory effort (thoracic and abdominal), body movement, and oxygen saturation were also taken. The measured variables included total sleep time, sleep efficiency (ratio between total sleep time and total recorded time multiplied by 100), sleep onset latency, wake after sleep onset, arousals, sleep stages (N1, N2 and N3 non-rapid eye movement [non-REM] sleep and REM sleep), latencies for each sleep stage. Two researchers who were blinded to the study design performed the staging and analysed the polysomnographic events using international criteria

SECONDARY OUTCOMES:
Change from baseline actigraphy sleep recording to first night and 6 weeks | baseline, first night, week 6
  It is an objective method to evaluate sleep by movement monitoring during the night. A wrist-watch-like package is used during at least one week. Measures include sleep onset latency, wakefulness after sleep onset, time in bed (TIB), total sleep time (TST), sleep efficiency (SE), and daytime napping. The device is used to assess sleep continuously during 10-day.
Change from baseline sleep diary recording to first night and 6 weeks | baseline, first night, week 6
  The sleep diary was used to evaluate the subjective perceptions of sleep. Participants were instructed to complete the diary every morning after waking for 10 days. The parameters evaluated were sleep onset latency, wake after sleep onset, total time in bed, number of arousals, sleep quality, feeling rested in the morning, and sleep efficiency (calculated retrospectively by the researchers as the ratio of reported total sleep time and reported total time in bed multiplied by 100). These data were averaged for each volunteer for pre- and post-treatment assessment weeks.
Change from baseline prior sleep anxiety to first night and 6 weeks | baseline, first night, week 6
  Prior sleep state anxiety will be assessed with the State-Trait Anxiety Inventory-STAI,25 the Portuguese version of which was validated by Gorenstein and Andrade.26 This scale encompasses 20 items and provides a one-dimensional measurement of anxiety. The volunteers were instructed to answer it 30 minutes before going to sleep at baseline and at the post-exercise evaluation.
Change from baseline insomnia severity to 12 weeks | baseline, week 6
  Insomnia Severity Index (ISI) was administrated at baseline and post treatment to assess insomnia-related complaints. It is a short and easy self-applied scale with 7 items scored from 0 to 4, with a total score varying from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia.
Change from baseline sleep quality to 6 weeks | baseline, week 6
  The PSQI assesses sleep quality over a 1-month period. The questionnaire consists of 19 self-rated questions and 5 questions that should be answered by bedmates or roommates. The latter questions are used only for clinical information. The 19 questions are categorized into 7 components, graded on a score that ranges from 0 to 3. The PSQI components are as follows: subjective sleep quality (C1), sleep latency (C2), sleep duration (C3), habitual sleep efficiency (C4), sleep disturbances (C5), use of sleeping medication (C6) and daytime dysfunction (C7). The sum of scores for these 7 components yields one global score, which ranges from 0 to 21, where the highest score indicates worst sleep quality. A global PSQI score greater than 5 indicates major difficulties in at least 2 components or moderate difficulties in more than 3 components.
Change from baseline mood to 6 weeks | baseline, week 6
  The POMS questionnaire is an instrument to evaluate the acute profile of mood. It has 65 items and 6 domains: tension-anxiety, depression, anger-hostility, vigour-activity, fatigue, and confusion- bewilderment. The total mood disturbance score is derived by subtracting the vigour-activity score from the the sum of scores from the other subscales.
Change from baseline quality of life to 6 weeks | baseline, week 6
  The SF-36 is a multidimensional questionnaire that covers eight components: physical functioning, role limitations due to physical health problems, role limitations due to emotional health problems, social functioning, vitality, general health perception, body pain, and mental health. All scores ranged from 0 to 100, with a higher score indicating better quality of life
Change from baseline serum serotonin to first night and 6 weeks | baseline, first night, week 6
  The serum serotonin dosage will be made by high performance liquid chromatography (HPLC). The blood sample will be collected at 8a.m.
Change from baseline cortisol to first night and 6 weeks | baseline, first night, week 6
  The cortisol dosage will be made by chemiluminescence. The blood sample will be collected at 8 a.m.
Change from baseline Effort Exercise test to 6 weeks | baseline, week 6
  The test will be performed on a treadmill according to the protocol of Bruce.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Padre Thiago, Jatai, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Undecided